CLINICAL TRIAL: NCT00135720
Title: A Double-Blinded, Placebo-Controlled Study of Etanercept (Enbrel) in the Treatment of Pemphigus Vulgaris
Brief Title: Study of Etanercept (Enbrel) in the Treatment of Pemphigus Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Stanford University (Other)
Responsible Party: Alexandra B. Kimball, Massachusetts General Hospital, Boston, MA 02114
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-P-002142; 79639;
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Pemphigus Vulgaris
Keywords: Pemphigus Vulgaris; Chronic Pemphigus; Etanercept; Enbrel; anti-TNF-alpha; TNF-alpha antagonist; biologic; immunomodulator; subcutaneous medication
MeSH Terms: conditions — Pemphigus | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Enbrel (Etanercept)

SUMMARY:
The purpose of the study is to find out about the effectiveness and the safety of an investigational drug called etanercept (Enbrel) to treat pemphigus vulgaris. Pemphigus vulgaris is a potentially life threatening blistering condition that currently has no cure.

An investigational drug is one that has not been approved by the United States (US) Food and Drug Administration (FDA) to treat a particular condition or disease. Etanercept has been approved by the FDA to treat rheumatoid arthritis, juvenile rheumatoid arthritis, and psoriasis, but not pemphigus vulgaris.

DETAILED DESCRIPTION:
People with pemphigus vulgaris have been found to have an increased amount of a substance called tumor-necrosis factor-alpha (TNF-alpha) in their blood. Etanercept may control pemphigus vulgaris by blocking the effect of TNF-alpha. Patients diagnosed with pemphigus vulgaris have been asked to participate in this research study.

Enrolled subjects will be given either etanercept or placebo. A placebo looks just like the study drug but contains no active medication. Placebos help study doctors find out if the effects of the study drug are due to the drug itself or just because of being in the study. This type of study design helps measure the true effectiveness of a treatment. Patients have 2 chances in 3 of receiving etanercept and 1 chance in 3 of receiving placebo.

The researchers expect to enroll 24 subjects in this study. Up to 16 subjects will be enrolled at Brigham and Women's Hospital (BWH) and Massachusetts General Hospital (MGH).

This study is sponsored by Amgen, Inc., the manufacturer of etanercept.

If taking part in another research study or have taken part in a research study in the last 28 days, patients will not be able to take part in this study. Patients cannot be on multiple studies simultaneously; however, exceptions are made for non-invasive, non-interventional, and observational studies.

This study will last about 16 weeks with a total of 6 study visits: screening, week 0 (baseline), weeks 2, 4, 8 and 16. The participants will be able to continue on your current medications for pemphigus throughout the study.

All participants must be at least 18 years of age with a clinical diagnosis of pemphigus vulgaris and at least 6 active blisters or erosions. Neither pregnant nor nursing women will be included in the study.

ELIGIBILITY:
Summary Inclusion Criteria:

* Understand and sign the written informed consent form and be willing and able to comply with the procedures of the study
* Have a clinical diagnosis of pemphigus vulgaris
* Have at least 6 active pemphigus lesions (blisters or erosions)
* Have no adverse effects due to combining etanercept with concurrent pemphigus medications
* Be on stable dose of current pemphigus medications for at least one month
* Females of child-bearing potential must have a negative urine pregnancy test prior to treatment and agree to practice an acceptable method of birth control (oral contraceptives, hormonal implant devices, Depo-Provera, condom with spermicide, diaphragm with contraceptive cream or foam, or intrauterine device) during the course of the study
* Be at least 18 years old at time of enrollment
* Be able to adhere to the study visit schedule and other protocol requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-06; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Determine the mean time (in days) it takes to reduce active lesions, including blisters and erosions, by 50%
Determine whether etanercept is a possible steroid-sparing treatment option. This will be determined by tapering the patient's existing steroid dose once our primary endpoint has been reached.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, MPH, Principal Investigator — CURTIS - Clinical Unit for Research Trials in Skin at Partners (MGH and BWH)
Locations (1):
- Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

REFERENCES:
- [Background] Stanley JR. Pemphigus. In Fizpatrick's Dermatology in General Medicine, 6th edition. Eds. Freedberg IM, Eisen AZ, Wolff K, Austen KF, et al. New York: McGraw-Hill, 2003. 558-567.
- [Background] Goldstein BG and Goldstein AO. Pemphigus and bullous pemphigoid. UpToDate.
- [Background] Alpsoy E, Yilmaz E, Basaran E, Yazar S, Cetin L. Is the combination of tetracycline and nicotinamide therapy alone effective in pemphigus? Arch Dermatol. 1995 Nov;131(11):1339-40. doi: 10.1001/archderm.131.11.1339. No abstract available. PMID 7503585
- [Background] Sacher C, Rubbert A, Konig C, Scharffetter-Kochanek K, Krieg T, Hunzelmann N. Treatment of recalcitrant cicatricial pemphigoid with the tumor necrosis factor alpha antagonist etanercept. J Am Acad Dermatol. 2002 Jan;46(1):113-5. doi: 10.1067/mjd.2001.119100. PMID 11756956
- [Background] Berookhim B, Fischer HD, Weinberg JM. Treatment of recalcitrant pemphigus vulgaris with the tumor necrosis factor alpha antagonist etanercept. Cutis. 2004 Oct;74(4):245-7. PMID 15551718
- [Background] Alecu M, Alecu S, Coman G, Galatescu E, Ursaciuc C. ICAM-1, ELAM-1, TNF-alpha and IL-6 in serum and blister liquid of pemphigus vulgaris patients. Roum Arch Microbiol Immunol. 1999 Apr-Jul;58(2):121-30. PMID 11845451
- [Background] D'Auria L, Bonifati C, Mussi A, D'Agosto G, De Simone C, Giacalone B, Ferraro C, Ameglio F. Cytokines in the sera of patients with pemphigus vulgaris: interleukin-6 and tumour necrosis factor-alpha levels are significantly increased as compared to healthy subjects and correlate with disease activity. Eur Cytokine Netw. 1997 Dec;8(4):383-7. PMID 9459618